CLINICAL TRIAL: NCT02910648
Title: Sleep Conditioning and Healthy Food Choices
Brief Title: Healthy Behaviors Learning Task and Sleep
Acronym: NAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00101818
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2021-08

CONDITIONS: Overweight/Obese Population
Keywords: healthy; BMI; weight loss; sleep; healthy sleeper; overweight; obese
MeSH Terms: conditions — Overweight; Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: We have adopted a randomized placebo control experimental design which requires the subjects to be blind to the subject's group assignment to minimize expectancy effects and the testing technician to be partially blind (blind to the sound cue group assignment and not blind to the go/no-go task) to minimize technician bias that could comprise the causal conclusions from being drawn.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Approach/Inhibit group (Experimental): Participants in the experimental group and control sham sound cues group will complete the Modified Go/No-Go Task.
  Following completion of post-training assessment measures, participants will be given the opportunity to take a 90-minute while undergoing real-time sleep monitoring.
  White noise will be played via headphones. Upon entering Stage N3 sleep and/or after having been asleep for 20 minutes and currently in any stage sleep other than N1, sound cues will be played to participants via headphones based on their randomization to 1 of 3 experimental groups.
  Interventions: Behavioral: Modified Go/No-Go Task
- Sham sound cues group (Sham Comparator): Participants in the experimental group and control sham sound cues group will complete the Modified Go/No-Go Task.
  Following completion of post-training assessment measures, participants will be given the opportunity to take a 90-minute while undergoing real-time sleep monitoring.
  White noise will be played via headphones. Upon entering Stage N3 sleep and/or after having been asleep for 20 minutes and currently in any stage sleep other than N1, sound cues will be played to participants via headphones based on their randomization to 1 of 3 experimental groups.
  Interventions: Behavioral: Modified Go/No-Go Task
- Sham go/no-go group (Sham Comparator): Participants in the control sham go/no-go group will complete a modified Go/No-Go Task with sham approach and inhibit items.
  Following completion of post-training assessment measures, participants will be given the opportunity to take a 90-minute while undergoing real-time sleep monitoring.
  White noise will be played via headphones. Upon entering Stage N3 sleep and/or after having been asleep for 20 minutes and currently in any stage sleep other than N1, sound cues will be played to participants via headphones based on their randomization to 1 of 3 experimental groups.
  Interventions: Behavioral: Modified Go/No-Go Task

INTERVENTIONS:
Behavioral: Modified Go/No-Go Task — Participants in the experimental group and control sham sound cues group will complete a computerized training task to facilitate learning to respond (press a computer key) to healthy food stimuli and to inhibit responses (not press a computer key) to unhealthy food stimuli. Participants in the control sham go/no-go group will complete a similar task with common office supplies (approach) and tools (inhibit). All participants will also complete a 24 hour dietary recall as described below.

SUMMARY:
This research is being done to study the impacts of a computerized learning task on health behaviors. The investigators are interested in studying whether this computerized learning task can help with weight loss.

DETAILED DESCRIPTION:
Over 1/3 of U.S. adults over the age of 20 are obese and obesity is associated with a host of deleterious medical comorbidities, including heart disease, type 2 diabetes, and cancer, costing the U.S. approximately $147 billion annually. Novel approaches to address this public health crisis are needed. Although obesity is multiply determined, it is ultimately a disorder of positive energy balance, such that weight loss requires increases in physical activity and improvements in choosing healthy over unhealthy foods. People who are strongly motivated to eat are more obese, and derive less benefit from weight loss treatments. There are two general approaches to addressing this pattern: 1) increase the reinforcing value of healthy foods and/or 2) increase an individual's self-control, i.e., the ability to inhibit approach responses to less healthy foods.

Emerging research has begun to develop and test training programs that directly modify tendencies to approach one type of stimulus while resisting temptation of another type of stimulus for problems other than obesity. For example, researchers have been able to train heavy drinkers to decrease their weekly alcohol intake7 and chocolate-lovers to reduce their chocolate intake. However, these researchers did not also incorporate increasing interest in alternatives (e.g., drinking water instead of beer). This training mechanism has also yet to be applied to research on obesity and decreasing intake of unhealthy foods.

Participants will be first trained via a computerized training task to inhibit responses to high-calorie (unhealthy) foods, and to approach alternative low-calorie, high-nutrient (healthy) foods, in order to test the tasks efficacy. The investigators will include the training task and incorporate a nap component consistent with Hu and colleagues to evaluate the utility of sleep conditioning for maintaining training-related changes in inhibition and approach tendencies after one week. Tones played during the training task will be played again during the nap, based on randomization

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 55, inclusive
* Body mass index ≥ 25
* Nonsmoker and non-nicotine user for a minimum of the past 6 months
* Not currently using recreational drugs
* Desire to lose weight
* Difficulty losing weight in the past
* AUDIT: <3 women, <4 men (note: score of 4 is okay if both items 2 and 3=0)
* Pittsburgh Sleep Quality Index questionnaire score <8
* Insomnia Severity Index questionnaire score <10
* Epworth Sleepiness Scale <10
* Below the clinical cutoff for Restless Leg Syndrome
* Full sleep cycle between 8:00pm and 9:00am at least 6 days per week
* Apnea hypopnea index <15, as measured by the Nox-T3

Exclusion Criteria:

* Current diagnosis of diabetes mellitus (type 1 or type 2)
* History of major medical disease impacting study
* Significant unstable medical morbidity within the past 6 months
* Significant unstable psychiatric disorder within the past 6 months
* Current use of antidepressants or opioids.
* Lifetime diagnosis of anorexia nervosa or bulimia nervosa
* Lifetime alcohol or substance abuse disorder or dependence
* Suicidal ideation in past year
* Lifetime serious head injury or stroke judged to impact pain or sleep
* Sleep disorder as assessed via the Structured Interview for sleep disorders (SIS-D).
* Women who are pregnant or lactating.
* Unwilling to follow study procedures
* Other (reason judged by PI)
* Food allergies: Individuals who report any food allergies or any history of anaphylactic reactions related to study procedures during the phone screen for this study will be excluded from participation. Participants who report avoidance of specific foods for other medical reasons (e.g., an interaction between a prescribed medication and a food group, food triggered migraines), if they are related to study procedures, will also be excluded from participation.
* Takes participant more than 30 minutes to fall asleep
* Positive toxicology screen

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2021-10-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Reinforcing Value of Food assessed by the Reinforcing Value of Food Questionnaire | Approximately 1 week (after second assessment has been taken)
  The reinforcing value of food task (RVF) assesses how hard an individual is willing to hypothetically work to gain access to food compared with an alternative. A series of paired-samples t-tests will be calculated in order to determine whether participants' scores on the reinforcing value of food test changed between baseline and 1 week later. Scores on the RVF have been shown to be associated with BMI. as well as obesity and energy intake.
Delay of Gratification assessed by the Kirby Questionnaire | Approximately 1 week (after second assessment has been taken)
  A series of paired-samples t-tests will be calculated in order to determine whether participants' scores on the Kirby Questionnaire changed between baseline and 1 week later. Each item is scored based on whether the participant chooses the shorter delay and less monetary reward versus the longer delay and a higher monetary reward. Delay-discounting rates are positively correlated with impulsiveness.
24 hour dietary recall: Nutrition Data System for Research (NDSR) assessed by the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) dietary food recall | Approximately 1 week (after second assessment has been taken)
  We will use paired-samples t-tests to determine whether participants mean caloric intake and macronutrient breakdown (e.g., %calories from fat) from the two dietary recalls pre-training task were significantly different from their means post-training task.
Go/no-go task assessed by the Go/no-go task | Approximately 1 week (after second assessment has been taken)
  Performance on go/no-go task as measured by reaction time and accuracy (combined into one score) will be correlated with baseline measures of dietary characteristics and disinhibition

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Smith, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Campus, Behavioral Medicine Research Lab, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No